CLINICAL TRIAL: NCT04148001
Title: Clinical and Laboratory Assessment Study of Patients With a Clinical Presentation Consistent With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: Identifying and Genotyping Homozygous Familial Hypercholesterolemia (HoFH) Patients
Status: Completed | Type: Observational
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-501-9101
Record Dates: First submitted 2019-10-11; First posted 2019-11-01 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Homozygous Familial Hypercholesterolemia (HoFH)
Keywords: LDL Receptors; Gene Therapy; Metabolic Diseases; Rare Diseases; Genetic Diseases; Atherosclerosis; Cardiovascular Disease; Genotype
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hyperlipoproteinemia Type II; Metabolic Diseases; Rare Diseases; Genetic Diseases, Inborn; Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Designed to help identify patients with HoFH due to mutations in the LDLR as confirmed by genotyping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to help identify patients with HoFH due to mutations in the LDLR as confirmed by genotyping.

DETAILED DESCRIPTION:
This is a non-interventional study; no investigational product is administered in this study. Information collected in this study may be used to identify potential participants for clinical gene therapy trials in HoFH.

The investigator will discuss the study with participants who have a clinical presentation consistent with HoFH and where possible, the treating physician, in order to assess their interest to participate. After informed consent has been obtained, participants will be asked to provide a blood sample (up to 40 mL) for genotyping to confirm genetic diagnosis of HoFH due to mutations in LDLR, a lipid panel and anti-AAV8 NAb titer. Participants and, whenever possible, their treating physician will complete a medical history questionnaire and provide supporting documentation. The informed consent form (ICF) and data collection methods may vary depending whether the informed consent is obtained remotely or at a participating study site.

Information collected will include the following:

* patient demographics (age, sex, weight)
* medical history
* previous genotype results (if available)
* results of most recent lipid panel(s)
* use of lipid lowering therapies, including failure to respond
* assessment of presence of liver disease, including history of hepatitis B and C, human immunodeficiency virus (HIV), cirrhosis, and alcohol use

Once this information is received by the investigator and Sponsor, a preliminary assessment of confirmation of a diagnosis of HoFH will be performed. Participants and/or their treating physician will be informed of the results of the genetic testing. All participants will be provided an opportunity to speak with a genetic counselor upon receiving the results of the genetic testing.

Data collected in this study may be used to identify potential candidates for separate clinical trial(s) using gene therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. Clinical presentation consistent with HoFH

Exclusion Criteria:

1. History of cirrhosis based on documented histological evaluation or noninvasive imaging
2. Documented diagnosis of liver diseases
3. History of immunodeficiency diseases, including a positive HIV test result
4. Previous organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females ≥ 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
The number of participants who have HoFH due to mutations in the LDLR gene measured by genetic testing | baseline
  The number of participants who have HoFH due to mutations in the LDLR (low density lipoprotein receptor) gene as confirmed by genetic testing.

SECONDARY OUTCOMES:
The measurement of AAV8 NAb titers | baseline
  The measurement of anti-AAV8 (adeno-associated virus serotype 8) neutralizing antibody (NAb) titers
The measurement of LDL-C, total cholesterol, very low density lipoprotein cholesterol (VLDL-C), non-high density lipoprotein cholesterol (non-HDL-C), high density lipoprotein cholesterol (HDL-C), triglycerides (TG), and lipoprotein a (Lp[a]) | baseline
  The measurement of LDL-C, total cholesterol, very low density lipoprotein cholesterol (VLDL-C), non-high density lipoprotein cholesterol (non-HDL-C), high density lipoprotein cholesterol (HDL-C), triglycerides (TG), and lipoprotein a (Lp[a]).
The number and types of the participant's current and historical lipid lowering therapies | baseline
  The number and types of lipid lowering therapies, including LDL-C apheresis, the participant has been on or is currently on
The participant's completion of the medical history questionnaire to determine relevant medical history | baseline
  Collection of the participant's relevant medical history

CONTACTS AND LOCATIONS:
Locations (1):
- Excel Medical Clinical Trials, LLC, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No